CLINICAL TRIAL: NCT06455878
Title: The Impact of Dietary Management Applet for Weight Reduction in Obese Heart Failure Patients: a Multicenter, Single-blind Randomized Controlled Trial
Brief Title: Mobile Applet for Weight Management in Obese Heart Failure Patients
Acronym: IDEAL-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Health Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Study2024-1
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Overweight and Obesity; Weight Loss; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full usage of diet management app group and with the full usage of an intelligent weight scale (Experimental): Full usage of the diet management app means subjects can use all functions of the application (including personal information, food record, weight record, exercise record, step count, daily dietary intake, distribution and analysis of dietary structure, and recommended foods and their structural distribution).
  Full usage of the intelligent weight scale means subjects can use all functions of the scale (including the report of heart rate, total body water, body fat rate, muscle mass, protein mass, bone mass, visceral fat index, basal metabolic rate, subcutaneous fat rate, and skeletal muscle rate).
  Interventions: Behavioral: Full usage of diet management app group and with the full usage of an intelligent weight scale
- Limited usage of diet management app group and with the limited usage of an intelligent weight scale (Active Comparator): Limited usage of the diet management app means subjects can use some functions of the application (including personal information, food record, weight record, exercise record, and step count).
  Limited usage of the intelligent weight scale means subjects can use a few functions of the scale (including the weight record, lower limb impedance value, and BMI).
  Interventions: Behavioral: Limited usage of diet management app group and with the limited usage of an intelligent weight scale

INTERVENTIONS:
Behavioral: Full usage of diet management app group and with the full usage of an intelligent weight scale — Subjects will use the fully functional diet management application and an intelligent weight scale with full function designed for obese heart failure patients to help them losed weight and invitigate some important composite cardiovascular endpoint.
  Arms: Full usage of diet management app group and with the full usage of an intelligent weight scale
Behavioral: Limited usage of diet management app group and with the limited usage of an intelligent weight scale — Subjects will use the limited function diet management application and an intelligent weight scale with limited function designed for obese heart failure patients as a comparator.
  Arms: Limited usage of diet management app group and with the limited usage of an intelligent weight scale

SUMMARY:
The objective of this clinical trial is to investigate the effect of weight reduction through a diet management application and an intelligent weight scale on a composite cardiovascular endpoint in obese patients with heart failure.

The main questions are:

Does the use of a diet management APP and intelligent weight scale reduce 1-year all-cause mortality, heart failure hospitalization, and first heart failure hospital stay? Does the use of a diet management APP and intelligent weight scale improve the outcomes of assessment of heart failure frailty and quality of life for heart failure?

Researchers will compare using the fully functional diet management app and intelligent weight scale to using the limitedly functional app and intelligent weight scale to see if the app works to improve heart failure conditions.

Participants will:

Use the diet management app at every meal and the intelligent weight scale every day for 12 months, and visit the clinic at 12 months for checkups.

DETAILED DESCRIPTION:
Obesity is one of the major risk factors for heart failure. Current guidelines for heart failure emphasize that severe obesity is associated with a poor prognosis in patients with heart failure, but there are no recommended effective interventions.

Caloric restriction alone, increased exercise, the use of weight-loss drugs, and bariatric surgery are not appropriate for obese patients with heart failure.

Whether obese heart failure patients with reduced ejection fraction (HFrEF) can benefit from weight loss treatment has not been evaluated in randomized controlled trials so far.

This study combines caloric restriction with lifestyle management to help HFrEF patients lose weight.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Left ventricular ejection fraction (LVEF) ≤ 50%, with New York Heart Association (NYHA) class II-III;
3. Body mass index (BMI) ≥ 26 kg/m² or male waist-to-hip ratio (WHR=waist circumference/hip circumference) ≥ 0.9, female waist-to-hip ratio ≥ 0.85;
4. Ability to use a smartphone and demonstrate compliance via a diet management mobile application during a 2-week ±1-week run-in period;
5. History of heart failure hospitalization within the past 6 months;
6. Signed informed consent.

Exclusion Criteria:

1. End-stage heart failure (≥2 hospitalizations for heart failure in the past 3 months, intolerance to guideline-directed medical therapy (GDMT), or dependence on inotropic agents);
2. Heart failure with reversible causes (e.g., peripartum cardiomyopathy, fulminant myocarditis);
3. Moderate or severe anemia (hemoglobin [Hb] <90 g/L);
4. Renal insufficiency (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m²) or ongoing dialysis;
5. Uncontrolled thyroid disease (hyperthyroidism/hypothyroidism) or end-stage liver failure;
6. Alcohol or substance abuse;
7. Current use of weight-loss medications or planned bariatric surgery;
8. Malignancy with an expected survival <1 year;
9. Conditions potentially hindering protocol compliance, as judged by the investigator (e.g., habitual reliance on food delivery services or company cafeteria meals);
10. Planned hospitalization during the trial period;
11. Concurrent participation in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hierarchical Composite Outcomes | Randomization through 1 year
  Patients experience "all-cause death, number of heart failure hospitalizations, time for the first heart failure hospitalization in days, assessment of heart failure frailty, heart failure-related quality of life, and percentage change of weight" by 1 year compared with baseline in the hierarchical composite endpoint analysis.
  Hierarchical composite outcome measure include:
  Death from any cause through 1 year; Number of hospitalizations due to heart failure through 1 year; Time for the first heart failure hospitalization in days through 1 year; Assessment of heart failure frailty (Fried Frailty Scale: score from 0 to 5, score ≥ 3 means frail, 1-2 means intermediate or pre-frail, 0 means robust); Heart failure-related quality of life (Kansas City Cardiomyopathy Questionnaire, KCCQ: score from 0 to 100, score 0-24 means quality of life is very poor to poor, 25-49 means poor to fair, 50-74 means fair to good, 75-100 means good to excellent); Percentage change of weight.

SECONDARY OUTCOMES:
Cardiovascular death within 1 year | From randomization to 1 year
  Events of Cardiovascular death happened
Number of heart failure hospitalizations within 1 year | From randomization to 1 year
  Number of hospitalizations due to heart failure through 1 year
Time of the first hospitalization for heart failure within 1 year | From randomization to 1 year
  The time of the first hospitalization in days for heart failure within 1 year
All cause death within 1 year | From randomization to 1 year
  Death from any cause through 1 year
Heart failure-related quality of life (KCCQ) | At baseline, 3-month and 1-year follow-ups.
  Heart failure-related quality of life (Kansas City Cardiomyopathy Questionnaire, KCCQ: score from 0 to 100; score 0-24 means quality of life is very poor to poor; 25-49 means poor to fair; 50-74 means fair to good; 75-100 means good to excellent).
Percentage change of weight | From randomization to 1 year
  Percentage change of weight compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rong Han, Study Director — Heart Health Research Center
Locations (26):
- China (26):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Langfang People's Hospital, Langfang, Hebei
  - Jixi City People's Hospital, Jixi, Heilongjiang
  - Luoyang No.6 People's Hospital, Luoyang, Henan
  - Ruyang County People's Hospital, Luoyang, Henan
  - Ningling County People's Hospital, Shangqiu, Henan
  - Yongcheng People's Hospital, Shangqiu, Henan
  - Shangcheng County People's Hospital, Xinyang, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Tongliao People's Hospital, Tongliao, Inner Mongolia
  - Xiu Yan Manchu Autonomous County Central People's Hospital, Anshan, Liaoning
  - Tiemei General Hospital of Liaoning Health Industry Group, Diaobingshancun, Liaoning
  - Shenyang Tenth Hospital, Shenyang, Liaoning
  - Pingdu People's Hospital, Pingdu, Shandong
  - Taian First Hospital, Taian, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Qin Yuan County People's Hospital, Changzhi, Shanxi
  - Xian Red Cross Hospital, Xian, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Yulin Branch Hospital, Yulin, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, The Xinjiang Uygur Autonomous Region
  - Yuhuan Second People's Hospital, Taizhou, Zhejiang
  - Beijing Chuiyangliu Hospital, Beijing
  - Beijing Fangshan District First Hospital, Beijing
  - Emergency General Hospital, Beijing
  - Kaifeng Central Hospital, Kaifeng

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam CSP, Gamble GD, Ling LH, Sim D, Leong KTG, Yeo PSD, Ong HY, Jaufeerally F, Ng TP, Cameron VA, Poppe K, Lund M, Devlin G, Troughton R, Richards AM, Doughty RN. Mortality associated with heart failure with preserved vs. reduced ejection fraction in a prospective international multi-ethnic cohort study. Eur Heart J. 2018 May 21;39(20):1770-1780. doi: 10.1093/eurheartj/ehy005. PMID 29390051
- [Background] Groenewegen A, Rutten FH, Mosterd A, Hoes AW. Epidemiology of heart failure. Eur J Heart Fail. 2020 Aug;22(8):1342-1356. doi: 10.1002/ejhf.1858. Epub 2020 Jun 1. PMID 32483830
- [Background] Aurigemma GP, de Simone G, Fitzgibbons TP. Cardiac remodeling in obesity. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):142-52. doi: 10.1161/CIRCIMAGING.111.964627. No abstract available. PMID 23322729
- [Background] Wang H, Li YY, Chai K, Zhang W, Li XL, Dong YG, Zhou JM, Huo Y, Yang JF. [Contemporary epidemiology and treatment of hospitalized heart failure patients in real clinical practice in China]. Zhonghua Xin Xue Guan Bing Za Zhi. 2019 Nov 24;47(11):865-874. doi: 10.3760/cma.j.issn.0253-3758.2019.11.004. Chinese. PMID 31744275
- [Background] Borlaug BA, Jensen MD, Kitzman DW, Lam CSP, Obokata M, Rider OJ. Obesity and heart failure with preserved ejection fraction: new insights and pathophysiological targets. Cardiovasc Res. 2023 Feb 3;118(18):3434-3450. doi: 10.1093/cvr/cvac120. PMID 35880317
- [Background] Koliaki C, Liatis S, Kokkinos A. Obesity and cardiovascular disease: revisiting an old relationship. Metabolism. 2019 Mar;92:98-107. doi: 10.1016/j.metabol.2018.10.011. Epub 2018 Nov 3. PMID 30399375
- [Background] Shariq OA, McKenzie TJ. Obesity-related hypertension: a review of pathophysiology, management, and the role of metabolic surgery. Gland Surg. 2020 Feb;9(1):80-93. doi: 10.21037/gs.2019.12.03. PMID 32206601
- [Background] Cao E, Watt MJ, Nowell CJ, Quach T, Simpson JS, De Melo Ferreira V, Agarwal S, Chu H, Srivastava A, Anderson D, Gracia G, Lam A, Segal G, Hong J, Hu L, Phang KL, Escott ABJ, Windsor JA, Phillips ARJ, Creek DJ, Harvey NL, Porter CJH, Trevaskis NL. Mesenteric lymphatic dysfunction promotes insulin resistance and represents a potential treatment target in obesity. Nat Metab. 2021 Sep;3(9):1175-1188. doi: 10.1038/s42255-021-00457-w. Epub 2021 Sep 20. PMID 34545251
- [Background] Kenchaiah S, Evans JC, Levy D, Wilson PW, Benjamin EJ, Larson MG, Kannel WB, Vasan RS. Obesity and the risk of heart failure. N Engl J Med. 2002 Aug 1;347(5):305-13. doi: 10.1056/NEJMoa020245. PMID 12151467
- [Background] Ho JE, Lyass A, Lee DS, Vasan RS, Kannel WB, Larson MG, Levy D. Predictors of new-onset heart failure: differences in preserved versus reduced ejection fraction. Circ Heart Fail. 2013 Mar;6(2):279-86. doi: 10.1161/CIRCHEARTFAILURE.112.972828. Epub 2012 Dec 27. PMID 23271790
- [Background] Brouwers FP, de Boer RA, van der Harst P, Voors AA, Gansevoort RT, Bakker SJ, Hillege HL, van Veldhuisen DJ, van Gilst WH. Incidence and epidemiology of new onset heart failure with preserved vs. reduced ejection fraction in a community-based cohort: 11-year follow-up of PREVEND. Eur Heart J. 2013 May;34(19):1424-31. doi: 10.1093/eurheartj/eht066. Epub 2013 Mar 6. PMID 23470495
- [Background] Pandey A, LaMonte M, Klein L, Ayers C, Psaty BM, Eaton CB, Allen NB, de Lemos JA, Carnethon M, Greenland P, Berry JD. Relationship Between Physical Activity, Body Mass Index, and Risk of Heart Failure. J Am Coll Cardiol. 2017 Mar 7;69(9):1129-1142. doi: 10.1016/j.jacc.2016.11.081. PMID 28254175
- [Background] Horwich TB, Fonarow GC, Clark AL. Obesity and the Obesity Paradox in Heart Failure. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):151-156. doi: 10.1016/j.pcad.2018.05.005. Epub 2018 May 28. PMID 29852198
- [Background] Butt JH, Petrie MC, Jhund PS, Sattar N, Desai AS, Kober L, Rouleau JL, Swedberg K, Zile MR, Solomon SD, Packer M, McMurray JJV. Anthropometric measures and adverse outcomes in heart failure with reduced ejection fraction: revisiting the obesity paradox. Eur Heart J. 2023 Apr 1;44(13):1136-1153. doi: 10.1093/eurheartj/ehad083. PMID 36944496
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e876-e894. doi: 10.1161/CIR.0000000000001062. Epub 2022 Apr 1. PMID 35363500
- [Background] Evangelista LS, Heber D, Li Z, Bowerman S, Hamilton MA, Fonarow GC. Reduced body weight and adiposity with a high-protein diet improves functional status, lipid profiles, glycemic control, and quality of life in patients with heart failure: a feasibility study. J Cardiovasc Nurs. 2009 May-Jun;24(3):207-15. doi: 10.1097/JCN.0b013e31819846b9. PMID 19390338
- [Background] Kitzman DW, Brubaker P, Morgan T, Haykowsky M, Hundley G, Kraus WE, Eggebeen J, Nicklas BJ. Effect of Caloric Restriction or Aerobic Exercise Training on Peak Oxygen Consumption and Quality of Life in Obese Older Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Jan 5;315(1):36-46. doi: 10.1001/jama.2015.17346. PMID 26746456
- [Background] Vest AR, Chan M, Deswal A, Givertz MM, Lekavich C, Lennie T, Litwin SE, Parsly L, Rodgers JE, Rich MW, Schulze PC, Slader A, Desai A. Nutrition, Obesity, and Cachexia in Patients With Heart Failure: A Consensus Statement from the Heart Failure Society of America Scientific Statements Committee. J Card Fail. 2019 May;25(5):380-400. doi: 10.1016/j.cardfail.2019.03.007. Epub 2019 Mar 13. PMID 30877038
- [Background] Margulies KB, Hernandez AF, Redfield MM, Givertz MM, Oliveira GH, Cole R, Mann DL, Whellan DJ, Kiernan MS, Felker GM, McNulty SE, Anstrom KJ, Shah MR, Braunwald E, Cappola TP; NHLBI Heart Failure Clinical Research Network. Effects of Liraglutide on Clinical Stability Among Patients With Advanced Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):500-8. doi: 10.1001/jama.2016.10260. PMID 27483064
- [Background] Jorsal A, Kistorp C, Holmager P, Tougaard RS, Nielsen R, Hanselmann A, Nilsson B, Moller JE, Hjort J, Rasmussen J, Boesgaard TW, Schou M, Videbaek L, Gustafsson I, Flyvbjerg A, Wiggers H, Tarnow L. Effect of liraglutide, a glucagon-like peptide-1 analogue, on left ventricular function in stable chronic heart failure patients with and without diabetes (LIVE)-a multicentre, double-blind, randomised, placebo-controlled trial. Eur J Heart Fail. 2017 Jan;19(1):69-77. doi: 10.1002/ejhf.657. Epub 2016 Oct 28. PMID 27790809
- [Background] Marso SP, Baeres FMM, Bain SC, Goldman B, Husain M, Nauck MA, Poulter NR, Pratley RE, Thomsen AB, Buse JB; LEADER Trial Investigators. Effects of Liraglutide on Cardiovascular Outcomes in Patients With Diabetes With or Without Heart Failure. J Am Coll Cardiol. 2020 Mar 17;75(10):1128-1141. doi: 10.1016/j.jacc.2019.12.063. PMID 32164886
- [Background] Bohula EA, Wiviott SD, McGuire DK, Inzucchi SE, Kuder J, Im K, Fanola CL, Qamar A, Brown C, Budaj A, Garcia-Castillo A, Gupta M, Leiter LA, Weissman NJ, White HD, Patel T, Francis B, Miao W, Perdomo C, Dhadda S, Bonaca MP, Ruff CT, Keech AC, Smith SR, Sabatine MS, Scirica BM; CAMELLIA-TIMI 61 Steering Committee and Investigators. Cardiovascular Safety of Lorcaserin in Overweight or Obese Patients. N Engl J Med. 2018 Sep 20;379(12):1107-1117. doi: 10.1056/NEJMoa1808721. Epub 2018 Aug 26. PMID 30145941
- [Background] Kosiborod MN, Abildstrom SZ, Borlaug BA, Butler J, Rasmussen S, Davies M, Hovingh GK, Kitzman DW, Lindegaard ML, Moller DV, Shah SJ, Treppendahl MB, Verma S, Abhayaratna W, Ahmed FZ, Chopra V, Ezekowitz J, Fu M, Ito H, Lelonek M, Melenovsky V, Merkely B, Nunez J, Perna E, Schou M, Senni M, Sharma K, Van der Meer P, von Lewinski D, Wolf D, Petrie MC; STEP-HFpEF Trial Committees and Investigators. Semaglutide in Patients with Heart Failure with Preserved Ejection Fraction and Obesity. N Engl J Med. 2023 Sep 21;389(12):1069-1084. doi: 10.1056/NEJMoa2306963. Epub 2023 Aug 25. PMID 37622681
- [Background] Berger S, Meyre P, Blum S, Aeschbacher S, Ruegg M, Briel M, Conen D. Bariatric surgery among patients with heart failure: a systematic review and meta-analysis. Open Heart. 2018 Dec 9;5(2):e000910. doi: 10.1136/openhrt-2018-000910. eCollection 2018. PMID 30613414
- [Background] Shimada YJ, Tsugawa Y, Brown DFM, Hasegawa K. Bariatric Surgery and Emergency Department Visits and Hospitalizations for Heart Failure Exacerbation: Population-Based, Self-Controlled Series. J Am Coll Cardiol. 2016 Mar 1;67(8):895-903. doi: 10.1016/j.jacc.2015.12.016. PMID 26916477
- [Background] Felker GM, Sharma A, Mentz RJ, She L, Green CL, Granger BB, Heitner JF, Cooper L, Teuteberg J, Grodin JL, Rosenfield K, Hudson L, Kwee LC, Ilkayeva O, Shah SH. A Randomized Controlled Trial of Mobile Health Intervention in Patients With Heart Failure and Diabetes. J Card Fail. 2022 Nov;28(11):1575-1583. doi: 10.1016/j.cardfail.2022.07.048. Epub 2022 Jul 23. PMID 35882260
- [Background] Dorsch MP, Farris KB, Rowell BE, Hummel SL, Koelling TM. The Effects of the ManageHF4Life Mobile App on Patients With Chronic Heart Failure: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 7;9(12):e26185. doi: 10.2196/26185. PMID 34878990